CLINICAL TRIAL: NCT01823666
Title: Study on Risk Factors for Prediction of Conversion to Dementia in Patients With Mild Cognitive Impairment
Brief Title: Predicting the Conversion From Mild Cognitive Impairment to Dementia
Acronym: PCMCItoD
Status: Completed | Type: Observational
Sponsor: Dongzhimen Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Jinzhou Tian, Professor, Dongzhimen Hospital, Beijing
Other Study IDs: Z11107056811043
Record Dates: First submitted 2013-03-30; First posted 2013-04-04 (Estimated); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Mild Cognitive Impairment; Alzheimer Disease; Dementia, Vascular
Keywords: Dementia; Alzheimer's disease; mild cognitive impairment
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease; Dementia, Vascular; Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Mild cognitive impairment: People with cognitive complaint will be recruited. Who can be diagnosed as mild cognitive impairment will be enrolled according to the MCI criteria.
- Control: Normal cognition.

SUMMARY:
Mild cognitive impairment (MCI) is believed to be the early stage of dementia. The investigators assume that some psychological and imaging risks may predict the conversion. In the current longitudinal study, psychological and imaging data of people with MCI will be obtained at baseline, and will be followed at 26 weeks and 52 weeks. The predictors will be found in comparison with controls.

DETAILED DESCRIPTION:
MCI increases the risk of later developing dementia. About 10-15% of the amnestic form of mild cognitive impairment will progress to Alzheimer's disease in one year. But some people with MCI never get worse. Others with MCI later have test results that return to normal for their age and education.

To develop a new drug for the prevention of dementia(dementia due to Alzheimer's disease or vascular dementia), investigators need a sensitive and specific tool for recognizing patients who will converse to dementia. The investigators want to establish an operational diagnostic criteria instead of a descriptive criteria for mild cognitive impairment.

ELIGIBILITY:
Inclusion Criteria:

* complaint about cognitive decline compared to previous performance
* objective cognitive impairment in one or more cognitive domains for age
* preservation of independence in functional abilities
* Mini-Mental State Examination(MMSE) scores between 24 and 30
* a Clinical Dementia Rating(CDR) score of 0.5

Exclusion Criteria:

* dementia
* patient with any following disease: Parkinson's disease, multiple system atrophy, normal pressure hydrocephalus, progressive supranuclear palsy, subarachnoid hemorrhage, brain neoplasms, Huntington disease, epilepsy
* depression(HAMD >7) or psychosis
* uncontrolled severe medical conditions(i.e., acute heart failure, renal insufficiency)
* current treatment with benzodiazepines, antidepressants, antipsychotics, or other medications with significant psychotropic or central cholinergic effects
* abnormal thyroid, low vitamin B12 level or low folic acid level
* patient with visual and auditory disorders can't cooperate with neuropsychological assessment
* patient can't cooperate with following up
* informed consent is not obtained

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with cognitive complaint living in the community.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2012-09; Primary Completion 2014-08 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Rate of conversion to dementia | At baseline, 26 weeks, and 52 weeks.

SECONDARY OUTCOMES:
Mini-Mental State Examination | At baseline, 26 weeks, and 52 weeks
Immediate and delayed story recall | At baseline, 26 weeks, and 52 weeks
Clock Drawing Test(CDT) | At baseline, 26 weeks, and 52 weeks
Boston Naming Test | At baseline, 26 weeks, and 52 weeks
Verbal Category Fluency Test(animals) | At baseline, 26 weeks, and 52 weeks
Trail Making Test(TMT) | At baseline, 26 weeks, and 52 weeks
Hopkins Verbal Learning Test(HVLT) | At baseline, 26 weeks, and 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jinzhou Tian, Doctor, Principal Investigator — Dongzhimen Hospital, Beijing
Locations (1):
- Dongzhimen Hospital affiliated to Beijing University of Chinese Medicine, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Ni J, Shi J, Wei M, Tian J, Jian W, Liu J, Liu T, Liu B. Screening mild cognitive impairment by delayed story recall and instrumental activities of daily living. Int J Geriatr Psychiatry. 2015 Aug;30(8):888-90. doi: 10.1002/gps.4317. No abstract available. PMID 26172064